CLINICAL TRIAL: NCT04381494
Title: Prospective, Interventional Pilot Study of Mobile Devices and Digital Applications to Detect Early Pneumonitis and Other Pulmonary Adverse Events in Unresectable Stage III Non-Small Cell Lung Cancer Patients on Durvalumab
Brief Title: Mobile Devices to Detect Early Pneumonitis in Stage III NSCLC Patients on Durvalumab.
Acronym: ON TRAX
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was not terminated for any safety concerns; it was stopped early due to inability to enroll patients in a timely manner and retain patients on study for the entire duration
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D4194C00008
Record Dates: First submitted 2020-04-02; First posted 2020-05-08 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-05

CONDITIONS: Unresectable Stage III NSCLC
Keywords: NSCLC; Non-Small Cell Lung Cancer; durvalumab; Stage III; Stage IIIA; Spirometer; Spirometry; PROs; Mobile Applications; Digital Applications; Stage IIIB; Stage IIIC; Device; Parametric; Pneumonitis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Observational/Other (Other): Patients will be enrolled after their treating physician has prescribed durvalumab and before they start durvalumab treatment. Patients will receive mobile and wearable devices alongside their durvalumab treatment without any additional interventions.
  Interventions: Device: Multiparametric Mobile Technology

INTERVENTIONS:
Device: Multiparametric Mobile Technology — Using a spirometer, an armband, and a tablet to collect data.

SUMMARY:
A study of whether mobile devices can improve the detection of pulmonary AEs (including pneumonitis) in stage III NSCLC patients post-CRT, while on durvalumab.

DETAILED DESCRIPTION:
Patients undergoing post-CRT treatment for lung cancer with consolidation durvalumab can experience pulmonary AEs that could become severe if not recognized and treated in time.

Data collected will be used to evaluate the likelihood of early detection of pulmonary AEs in unresectable Stage III NSCLC patients on durvalumab. This project seeks to understand if multiparametric mobile technology collecting patient reported outcomes, vital signs, and respiratory function, integrate well into a patients daily life and aid physicians in early detection of pulmonary AEs.

ELIGIBILITY:
Select Inclusion Criteria:

* Patient has unresectable Stage III NSCLC that has not progressed following concurrent platinum-based chemotherapy and radiation therapy and is eligible to receive durvalumab according to the US FDA approved package insert.
* Patient is able and willing to use the mobile application and connected devices.
* Patient is able to complete QoL assessments.

Select Exclusion Criteria:

* Patient is currently oxygen dependent.
* Patient has comorbidities that will prevent consistent and reliable measurement assessments with multiparametric mobile technology including severe chronic obstructive pulmonary disorder (COPD), severe asthma, congestive heart failure [CHF], interstitial lung disease [ILD], and others.
* Patients on other immunotherapy or systemic immunosuppressants.
* Patients with active or prior autoimmune disease or history of immunodeficiency.
* Currently pregnant women.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Research Site, Long Beach, California
  - Research Site, Santa Ana, California
  - Research Site, Englewood, Colorado
  - Research Site, Plainville, Connecticut
  - Research Site, Boca Raton, Florida
  - Research Site, Tallahassee, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Westwood, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, Pontiac, Michigan
  - Research Site, New York, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Massillon, Ohio
  - Research Site, Knoxville, Tennessee
  - Research Site, San Antonio, Texas
  - Research Site, Lacey, Washington
  - Research Site, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4194C00008&attachmentIdentifier=7035ee52-a3a7-4c19-a4bf-70642e355403&fileName=D4194C00008_Protocol_Redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4194C00008&attachmentIdentifier=2138fa46-a8da-4441-97a2-eceaeb1c7369&fileName=D4194C00008_SAP_Redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4194C00008&attachmentIdentifier=42b0fdcc-82c1-46ab-b2a4-e0a31e0c5758&fileName=D4194C00008-CSR_Synopsis.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a prospective, interventional pilot study of mobile devices and digital applications conducted at 25 sites in the United States to detect early signs of pneumonitis and other pulmonary adverse events (AEs) in participants with unresectable Stage III Non-Small Cell Lung Cancer (NSCLC) whose disease had not progressed following 2 or more cycles of concurrent chemoradiotherapy, treated with durvalumab.
Pre-assignment Details: A total of 40 participants were enrolled in this study after their treating physician prescribed durvalumab and before starting durvalumab. Data was collected via Current Wearable Health Monitoring System.
Groups:
- All Participants: Participants were trained on the mobile applications and received mobile and wearable devices alongside their durvalumab treatment without any additional interventions. Participants received durvalumab for up to 12 months or until confirmed disease progression, permanent discontinuation of durvalumab, the initiation of alternative cancer therapy, unacceptable toxic events, death, or withdrawal of consent, whichever was sooner.
Period: Overall Study
Arm/Group | All Participants
Started | 40
Completed | 5
Not Completed | 35
Not completed — Early termination of trial | 19
Not completed — Investigator's discretion | 1
Not completed — Withdrawal by Subject | 9
Not completed — NSCLC disease progression | 4
Not completed — Device-Related Adverse Event | 2

BASELINE CHARACTERISTICS:
Population: The Safety Analysis set (SAF) included all enrolled participants who took at least 1 dose of durvalumab.
Arm/Group | All Participants
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (8.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Event (TEAE) of Pneumonitis by Grade
Description: An AE was occurrence of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product or device, whether or not considered causally related to the product or device medical occurrence in a participant. The TEAEs of pneumonitis were defined as any pneumonitis event that occurred or worsened at any time after the start of administration of the first dose of durvalumab and through 30 days after the last dose of durvalumab. Severity (intensity of any event) was assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse events (CTCAE) v5. The AEs were assigned to a Grade from 1 through 5 as follows: Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe or medically significant but not immediately life-threatening requiring hospitalization; Grade 4: Life-threatening consequences; Grade 5: Death due to any AE.
Time Frame: TEAEs were reported from the first dose of durvalumab up to 30 days after the last dose of durvalumab, a maximum of approximately 13 months
Population: The SAF included all enrolled participants who took at least 1 dose of durvalumab.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 40
Participants
  Grade 2 | 2
  Grade 3 | 1

2. Secondary Outcome: Number of Participants With Permanent Discontinuation of Durvalumab Due to Pulmonary TEAEs
Description: Pulmonary TEAEs were defined as any pulmonary AEs that occurred or worsened at any time after the start of administration of the first dose of durvalumab and through 30 days after the last dose of durvalumab. Number of participants with permanent discontinuation of durvalumab due to pulmonary TEAEs including pneumonitis are reported.
Time Frame: as for outcome 1
Population: The SAF included all enrolled participants who took at least 1 dose of durvalumab.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 40
Participants | 0

3. Secondary Outcome: Duration of Durvalumab Treatment
Description: The overall duration of durvalumab treatment, while participants were a part of this wearable study, was calculated as end date of durvalumab treatment minus first dose of durvalumab (Day 1) plus 1.
Time Frame: Up to Month 12
Population: The SAF included all enrolled participants who took at least 1 dose of durvalumab.
Measure: Mean (Full Range); unit: days
Arm/Group | All Participants
Number analyzed (Participants) | 40
days | 107.5 [1 to 352]

4. Secondary Outcome: Number of Participants With Early Discontinuation of Durvalumab
Description: Number of participants who discontinued durvalumab early due to any reason are reported.
Time Frame: Up to Month 12
Population: The SAF included all enrolled participants who took at least 1 dose of durvalumab.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 40
Participants | 3

5. Secondary Outcome: Number of Participants With Treatment Interruptions
Description: Treatment interruptions were defined as at least 1 temporary withholding of durvalumab treatment. Treatment withheld was defined as temporarily withheld of durvalumab recorded in case report form. Short interruptions defined as the durvalumab infusion interruption during the administration recorded in CRF in a single visit were excluded from the analysis. Due to data issue, the reason for treatment withheld was not captured in the database.
Time Frame: Up to Month 12
Population: The SAF included all enrolled participants who took at least 1 dose of durvalumab.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 40
Participants | 9

6. Secondary Outcome: Duration of Durvalumab Treatment Interruption
Description: The overall duration of durvalumab treatment interruption was calculated as the sum of the duration of each treatment withheld/resumed. The duration of interruption included only treatment withheld. Short interruption which resumed during the same visit was not included in the calculation for duration of interruption.
Time Frame: Up to Month 12
Population: The SAF included all enrolled participants who took at least 1 dose of durvalumab.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | All Participants
Number analyzed (Participants) | 40
days | 50.8 (50.79)

7. Secondary Outcome: Number of Participants With Pulmonary TEAEs Excluding Pneumonitis
Description: Pulmonary TEAEs were defined as any pulmonary AEs that occurred or worsened at any time after the start of administration of the first dose of durvalumab and through 30 days after the last dose of durvalumab.
Time Frame: as for outcome 1
Population: The SAF included all enrolled participants who took at least 1 dose of durvalumab.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 40
Participants | 19

8. Secondary Outcome: Duration of Pulmonary TEAEs Excluding Pneumonitis
Description: Pulmonary TEAEs were defined as any pulmonary AEs that occurred or worsened at any time after the start of administration of the first dose of durvalumab and through 30 days after the last dose of durvalumab. Duration of pulmonary TEAEs was calculated as end date of pulmonary TEAE minus onset date of pulmonary TEAE plus 1. For AEs that were missing an end date, the data cut-off date was used as the AE end date for calculation of AE duration.
Time Frame: as for outcome 1
Population: The SAF included all enrolled participants who took at least 1 dose of durvalumab. Only those participants with pulmonary TEAEs excluding pneumonitis were included in this analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | All Participants
Number analyzed (Participants) | 19
days | 153.4 (156.26)

9. Secondary Outcome: Number of Participants Who Received Prescription Medication to Manage Pneumonitis TEAEs
Description: Pneumonitis TEAEs were defined as any pneumonitis AEs that occurred or worsened at any time after the start of administration of the first dose of durvalumab and through 30 days after the last dose of durvalumab.
Time Frame: Up to Month 12
Population: The SAF included all enrolled participants who took at least 1 dose of durvalumab. Only those participants with pneumonitis TEAEs were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 3
Participants | 2

10. Secondary Outcome: Duration of Prescription Medication Received by Participants to Manage Pneumonitis TEAEs
Description: as for outcome 9
Time Frame: Up to Month 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: days
Arm/Group | All Participants
Number analyzed (Participants) | 2
days | 17.5 (3.54)

11. Secondary Outcome: Duration of Development of Grade 3 to Grade 5 TEAEs, Including Pneumonitis
Description: Duration of development of Grade 3 to 5 pneumonitis AEs is defined as the period from Day 1 to earliest of each grade of pneumonitis AE (grade 3, grade 4, and grade 5). Severity (intensity of an event) was assessed using the NCI-CTCAE v5. AEs were assigned to a Grade from 1 through 5 as follows: Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe or medically significant but not immediately life-threatening requiring hospitalization; Grade 4: Life-threatening consequences; Grade 5: Death due to any AE.
Time Frame: as for outcome 1
Population: Data was not collected due to early termination of the trial.
Arm/Group | All Participants
Number analyzed (Participants) | 0

12. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 Items (EORTC QLQ-C30) in Participants With Pneumonitis TEAEs
Description: The EORTC QLQ-C30 consisted of 30 questions and included functional scales (FS) (items 1-7 and items 20-27), symptom scales (items 8-19 and item 28) and global measure of health status (GHS) (items 29-30). The scale ranged from 1-4 for most outcome measures of systems, with 1 rated as "not at all" and 4 rated as "very much". Scores were averaged and transformed to 0 to 100, a high score for functional scales/GHS represented better functioning ability/QoL, whereas a high score for symptom scales represented stronger symptoms/worse QoL. Participants with pneumonitis TEAEs with causal relationship with durvalumab are presented. Time point 1: prior to occurrence of initial pneumonitis AE; Time point 2: at same time point as initial pneumonitis AE; Time point 3: when highest CTCAE grade of pneumonitis AE occurred. Baseline was defined as the date of informed consent for this parameter.
Time Frame: Baseline visit (Day 1), every 2 weeks for the first 3 months and once monthly thereafter, and at End-of-Study visit (Month 12)
Population: The SAF included all enrolled participants who took at least 1 dose of durvalumab. For each symptom scale, only those participants with data available were included in the analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 40
scores on a scale
  FS; Time point 1: number analyzed (Participants) | 2
  FS; Time point 1 | 5.56 (4.714)
  FS; Time point 2: number analyzed (Participants) | 1
  FS; Time point 2 | 2.22 (NA) — Standard deviation could not be calculated for single participant.
  FS; Time point 3: number analyzed (Participants) | 1
  FS; Time point 3 | 2.22 (NA) — Standard deviation could not be calculated for single participant.
  Symptom scale; Time point 1: number analyzed (Participants) | 2
  Symptom scale; Time point 1 | -10.26 (3.626)
  Symptom scale; Time point 2: number analyzed (Participants) | 1
  Symptom scale; Time point 2 | -7.69 (NA) — Standard deviation could not be calculated for single participant.
  Symptom scale; Time point 3: number analyzed (Participants) | 1
  Symptom scale; Time point 3 | -7.69 (NA) — Standard deviation could not be calculated for single participant.
  GHS; Time point 1: number analyzed (Participants) | 2
  GHS; Time point 1 | 4.17 (5.893)
  GHS; Time point 2: number analyzed (Participants) | 1
  GHS; Time point 2 | 8.33 (NA) — Standard deviation could not be calculated for single participant.
  GHS; Time point 3: number analyzed (Participants) | 1
  GHS; Time point 3 | 8.33 (NA) — Standard deviation could not be calculated for single participant.

13. Secondary Outcome: Change From Baseline in EORTC QLQ-Lung Cancer (LC)13 in Participants With Pneumonitis TEAEs
Description: The EORTC QLQ-LC13 was a disease-specific 13-item questionnaire for lung cancer used in conjunction with the EORTC QLQ-C30. It comprised both multi-item and single-item measures of lung cancer associated symptoms (LCAS) (items 31-35 and items 40-42), treatment related side effects (TREF) (items 36-39) and pain medication (item 43). The scale ranged from 1-4 for most outcome measures of systems, 1 rated as "not at all" and 4 rated as "very much". Scores were averaged and transformed to 0 to 100, higher scores for LCAS and TREF: greater level of symptoms/worse QoL and higher scores for pain medication: better pain relief from medication. Participants with pneumonitis TEAEs with causal relationship with durvalumab are presented. Time point 1: prior to occurrence of initial pneumonitis AE; Time point 2: at same time point as initial pneumonitis AE; Time point 3: when highest CTCAE grade of pneumonitis AE occurred. Baseline was defined as the date of informed consent for this parameter.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 40
scores on a scale
  LCAS; Time point 1: number analyzed (Participants) | 1
  LCAS; Time point 1 | -4.17 (NA) — Standard deviation could not be calculated for single participant.
  LCAS; Time point 2: number analyzed (Participants) | 0
  LCAS; Time point 3: number analyzed (Participants) | 0
  TREF; Time point 1: number analyzed (Participants) | 1
  TREF; Time point 1 | -8.33 (NA) — Standard deviation could not be calculated for single participant.
  TREF; Time point 2: number analyzed (Participants) | 0
  TREF; Time point 3: number analyzed (Participants) | 0
  Pain medication; Time point 1: number analyzed (Participants) | 1
  Pain medication; Time point 1 | 0 (NA) — Standard deviation could not be calculated for single participant.
  Pain medication; Time point 2: number analyzed (Participants) | 0
  Pain medication; Time point 3: number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: TEAEs were reported from the first dose of durvalumab up to 30 days after the last dose of durvalumab, a maximum of approximately 13 months
Description: The SAF included all enrolled participants who took at least 1 dose of durvalumab.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 1/40
Serious Adverse Events (participants affected / at risk) | 5/40
Other Adverse Events (participants affected / at risk) | 20/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=40)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=40)
Diarrhoea (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 4 (6)
Fatigue (General disorders) | 7 (8)
Non-cardiac chest pain (General disorders) | 4 (4)
Pyrexia (General disorders) | 5 (5)
Tachycardia (Cardiac disorders) | 4 (4)
Dizziness (Nervous system disorders) | 4 (6)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (4)

LIMITATIONS AND CAVEATS:
This pilot trial was terminated early due to the Coronavirus Disease-2019 (COVID-19) pandemic, shortage of site staff, and limited access to sites resulting in participant enrollment and retention challenges. The trial was not terminated early due to any safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-12-02): https://cdn.clinicaltrials.gov/large-docs/94/NCT04381494/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/94/NCT04381494/SAP_001.pdf